CLINICAL TRIAL: NCT07299266
Title: Doctoral Thesis Study
Brief Title: The Impact of Mobile Application-Supported Monitoring on Treatment Compliance and Success in Lifestyle Changes in Hypertensive Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Mehmet Ali Bozkurt, PhD Student, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/140
Record Dates: First submitted 2025-11-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This study was planned as a randomized, controlled and experimental study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Mobile App-Supported Follow-Up (Experimental): Participants in this group will be provided with a Bluetooth-enabled digital blood pressure device and an integrated mobile application. Following the pre-test administration, participants in the intervention group will be provided with a digital blood pressure monitoring device featuring Bluetooth synchronization, and an integrated mobile application will be installed on their smartphones. Blood pressure measurements taken by the participants will be automatically recorded via the mobile application and stored in a digital database. Furthermore, the application will send regular automated reminders and notifications to participants regarding:
  Medication intake times
  Physician follow-up appointments
  Periodic blood pressure measurement times
  This intervention aims to facilitate technology-supported monitoring and proactive patient management.
  Interventions: Behavioral: Mobile App-Supported Blood Pressure Monitoring
- Control Group - Standard Follow-Up (No Intervention): Participants in the control group will be provided with a standard digital blood pressure monitoring device that does not have Bluetooth capability. These participants will be instructed to perform their blood pressure measurements regularly and to manually record them on the printed follow-up forms provided to them. The control group will not receive the additional technological support offered to the intervention group, such as the mobile application, automatic data recording, and reminder system; instead, the standard follow-up process will be observed.

INTERVENTIONS:
Behavioral: Mobile App-Supported Blood Pressure Monitoring — Participants will be provided with a Bluetooth-enabled digital blood pressure device integrated with a mobile application. The application will automatically record blood pressure measurements and provide automated reminders for medication intake, scheduled blood pressure measurements, and follow-up appointments. This intervention aims to enhance treatment adherence and promote successful lifestyle modifications in patients with hypertension.
  Arms: Intervention Group - Mobile App-Supported Follow-Up

SUMMARY:
Hypertension (HT) is defined as an arterial blood pressure persistently exceeding 140/90 mmHg in repeated measurements. It is a systemic disease characterized by chronically elevated blood pressure, which can lead to severe health complications. Despite advancements in screening, diagnosis, and treatment methods, hypertension remains a leading risk factor for mortality and disability in both developed and developing countries. Globally, approximately 1.3 billion individuals are living with hypertension. It is projected that within the next two decades, hypertension will become the most significant modifiable risk factor for non-communicable diseases. International guidelines recommend ambulatory blood pressure monitoring (ABPM) and/or home blood pressure monitoring (HBPM) for the diagnosis of hypertension. It has been demonstrated that home and/or ambulatory blood pressure measurements provide superior prognostic information regarding target organ damage and cardiovascular risk compared to clinic-based measurements. Nevertheless, both ambulatory and home blood pressure monitoring have several well-known limitations, including patient comfort, sleep disturbance, accessibility, and cost.

The use of various mobile technologies has been evaluated in different settings to improve hypertension management in primary care services. Mobile monitoring can lead to significant reductions in blood pressure (BP), decrease all-cause and hypertension-related hospitalizations, lower all-cause mortality and costs, and enhance quality of life. Furthermore, technology-assisted BP self-monitoring interventions have demonstrated superior BP control outcomes when combined with nurse-led mobile support, physician intervention, and medication review. This research, grounded in the integration of digital health technologies into nursing care, aims to enhance treatment adherence and the success of lifestyle modifications in hypertensive patients through mobile application-supported monitoring. Through this approach, the patient-nurse interaction will be strengthened, and self-management skills will be supported via personalized feedback.

DETAILED DESCRIPTION:
1. Research Design/Model/Type:

   Method of the study: This study is planned as randomized, controlled and experimental. Study Population and Sample The study population will consist of hypertensive patients who are under follow-up at the cardiology and internal medicine outpatient clinics of Kilis Prof. Dr. Alaeddin Yavaşca State Hospital. The sample will be composed of patients diagnosed with Hypertension (HT) who meet the inclusion criteria, with the sample size determined through a power analysis. Participants will be assigned to either an intervention or a control group using a simple random sampling method.

   Intervention and Control Groups Participants in the intervention group will be provided with a digital blood pressure monitoring device with Bluetooth capability and a mobile application that integrates with this device. Measurements taken by the participants will be automatically recorded via the mobile application. Furthermore, the application will provide automated reminders for medication intake, scheduled blood pressure measurements, and follow-up appointments.

   Participants in the control group will be given a standard digital blood pressure device without Bluetooth functionality, and their measurements will be stored in the device's internal memory. The control group will not receive any additional technological support, such as a mobile application or digital reminders.

   Study Setting and Duration The study will be conducted at the cardiology and internal medicine outpatient clinics of Kilis Prof. Dr. Alaeddin Yavaşca State Hospital. The data collection process will commence after receiving the necessary approvals from the ethics committee and the institution. The total planned duration of the study is 18 months, which includes the phases of preliminary preparation, data collection, a three-month follow-up period, and analysis.
2. Study Group/Sample of the Study: The sample of this study will consist of a total of 40 patients, including 20 in the intervention group and 20 in the control group, as calculated based on a power analysis.

   In the power analysis, the study by Chandler et al. (2019) titled "Impact of a culturally tailored mHealth medication regimen self-management program upon blood pressure among hypertensive Hispanic adults" was used as a reference. According to this study, assuming a large effect size (d = 0.92) between the treatment adherence scores of the group using the mobile application and the group not using it, the minimum required sample size was determined as 20 participants per group to achieve statistical significance at α = 0.05 and power (1-β) = 0.80.

   The power analysis was conducted using the G*Power 3.9.1 software with the following parameters:

   t tests - Means: Difference between two independent means (two groups). Analysis: A priori: Compute required sample size. Input: Tail(s) = Two; Effect size d = 0.9216752; α err prob = 0.05; Power (1-β err prob) = 0.80; Allocation ratio N2/N1 = 1.

   Output: Noncentrality parameter δ = 2.9145929; Critical t = 2.0243942; df = 38; Sample size group 1 = 20; Sample size group 2 = 20; Total sample size = 40; Actual power = 0.8106404.
3. Data Collection Tools to be Used in the Project/Research:

   1. Question Form: Data will be collected from the patients through face-to-face interviews using a questionnaire developed by the researchers. This form was designed to gather the participants' demographic and clinical characteristics, such as age, gender, marital status, educational level, occupation, duration of illness, and medication use. The questionnaire consists of 42 items and was created by the researchers based on a review of the relevant literature.
   2. Evaluation Scale for Treatment Compliance and Life Change Success of Hypertensive Individuals: The levels of treatment adherence and lifestyle modification success among patients will be measured using the "Scale for Assessing Treatment Adherence and Lifestyle Modification Success in Hypertensive Individuals." The scale is composed of 18 items and consists of five factors. Items on the scale are scored on a five-point Likert scale ranging from "Never" (1 point) to "Always" (5 points), with intermediate anchors of "Rarely" (2 points), "Sometimes" (3 points), and "Frequently" (4 points).

The scale has five sub-dimensions:

Adherence to medical treatment (items 1, 2, 3, 4, 5) Communication with the physician during the treatment process (items 13, 14, 15) Healthy diet (items 7, 8, 9) Physical activity and weight control (items 10, 11, 12) Salt and processed food consumption (items 16, 17, 18) The total score obtainable from the scale ranges from 18 to 90. The optimal cut-off point for the scale, determined by the ROC curve method, has been established at 68 points.

c. Study Procedure Prior to the commencement of the study, participants will be informed about the research, and their written and verbal consent will be obtained. At the beginning of the study, the Questionnaire Form and the "Scale for Assessing Treatment Adherence and Lifestyle Modification Success in Hypertensive Individuals" will be administered as a pre-test to all participants in both groups.

Procedure for the Intervention Group

Following the pre-test administration, participants in the intervention group will be provided with a digital blood pressure monitoring device featuring Bluetooth synchronization, and an integrated mobile application will be installed on their smartphones. Blood pressure measurements taken by the participants will be automatically recorded via the mobile application and stored in a digital database. Additionally, the mobile application will send regular automated reminders and notifications to the participants regarding:

* Medication intake times
* Physician follow-up appointments
* Periodic blood pressure measurement times

This intervention aims to provide technology-supported monitoring and proactive patient management.

Procedure for the Control Group Participants in the control group will be given a standard digital blood pressure monitoring device without Bluetooth capability. These participants will be instructed to perform their blood pressure measurements regularly and to manually record them on printed follow-up forms provided to them. The control group will not receive the additional technological support offered to the intervention group, such as the mobile application, automatic data recording, or the reminder system; they will follow the standard care protocol.

At the conclusion of the specified follow-up period, the same measurement instruments administered at the beginning will be re-administered as a post-test to both groups. The effectiveness of the intervention will then be evaluated through an inter-group comparison. This methodology will allow for the examination of the efficacy of the mobile health-based monitoring intervention on patients' clinical parameters and treatment adherence compared to standard care.

d. Evaluation of Project/Research Data: Data will be evaluated using the Statistical Package for Social Sciences-SPSS 25.0 package program, and frequency, percentage, mean and standard deviation will be used as descriptive statistics, and Shapiro Wilk test will be used to check the normal distribution of continuous variables. Student t, Chi-square, Mann-Whitney U and Kruskal Wallis, Anova tests will be applied under appropriate conditions to examine the differences between categorical variables. The statistical significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hypertension at least 6 months prior.
* Willingness to voluntarily participate in the study.
* Aged 18 years or older.
* Ability to use a smartphone.
* Ability to read and write (literate).

Exclusion Criteria:

* Patients with other serious cardiovascular diseases (e.g., heart failure, cardiac arrhythmia).
* Inability to use a smartphone (for the intervention group).
* Pregnancy.
* Withdrawal of consent or request to leave the study.
* Presence of any diagnosed psychiatric disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Systolic and Diastolic Blood Pressure at Month 3 | Baseline, Month 3 (3 months)
  Participants' blood pressure will be measured twice daily (morning and evening) for 3 months. In the intervention group, measurements are automatically transferred to a mobile application via Bluetooth-enabled devices. In the control group, measurements are recorded in the memory of standard digital devices. Results are reported in millimeters of mercury (mmHg). The change in mean blood pressure values between baseline and the end of Month 3 will be analyzed.
Change from Baseline in "Scale for Assessment of Treatment Adherence and Lifestyle Change Success in Hypertensive Individuals" Total Score at Month 3 | Baseline and Month 3
  Treatment adherence and lifestyle changes will be assessed using the "Scale for Assessment of Treatment Adherence and Lifestyle Change Success in Hypertensive Individuals" (Hipertansif Bireylerin Tedaviye Uyum ve Yaşam Değişikliği Başarısını Değerlendirme Ölçeği) developed by Esirgen (2018). The scale consists of 18 items across 5 sub-dimensions (medical treatment adherence, communication with physician, healthy nutrition, physical activity and weight control, and salt and fast food consumption). The total score ranges from 18 (minimum) to 90 (maximum). Higher scores indicate better treatment adherence and positive lifestyle behaviors; a score of 68 or higher is considered "compliant". The change in the total score between baseline and the end of Month 3 will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ovayolu, Prof. Dr., Study Director — https://www.gaziantep.edu.tr/

IPD SHARING:
Plan to Share IPD: No
The research data will remain confidential by the researchers.